CLINICAL TRIAL: NCT05370586
Title: Pericapsular Nerve Group (PENG) Block Versus Fascia Iliaca (FIB) Block for Emergency Department Analgesia in Hip Fractures: A Randomised Controlled Trial.
Brief Title: PENG Block vs Fascia Iliaca Block for Emergency Department Analgesia in Hip Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Colchester General Hospital (Other)
Responsible Party: Principal Investigator, Santi Di Pietro, MD, PhD - Emergency Medicine Consultant, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0020199/22
Record Dates: First submitted 2022-05-07; First posted 2022-05-11 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Hip Fractures
Keywords: Fascia iliaca block; PENG block; Regional anaesthesia at Emergency Departments; Hip Fracture Analgesia
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: andomised-controlled trial with two parallel study groups. Participants will be randomised 1:1 to the study or control group. The study group will be treated with PENG block following randomisation, whereas the control group will receive the standard treatment, i.e., fascia iliaca block.
  The study aims to demonstrate the superiority of the new intervention over the standard approach.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG block: Study group (Experimental): Patients enrolled in the study group will receive a PENG block with 20 mL of 0,375% levobupivacaine with 4 mg of dexamethasone. The block will be performed with the patient in a supine position using an 18-gauge, 90 mm needle, inserted with an in-plane lateral to medial approach. Operators will use the original technique described by Girón-Arango L et al. The aim of this block is to inject the local anaesthetic between the psoas tendon and the iliopubic eminence. We will instruct operators to routinely use a curvilinear probe (2-6 MHz) or a linear probe (4-16 MHz) in particularly lean or cachectic patients.
  Interventions: Other: Pericapsular nerve Group Block
- Infrainguinal fascia iliaca block: Control group (Other): Patients allocated in the control group will receive an infrainguinal fascia iliaca block with 30 mL of 0,25 % levobupivacaine with 4 mg of dexamethasone, using an 18-gauge, 90 mm needle, inserted with an in-plane lateral to medial approach.
  The probe (linear 4-16 MHz) is placed transversely at the inguinal crease to identify the femoral artery, femoral nerve, iliopsoas muscle and the fascia iliaca over the psoas muscle. Moving the probe laterally the sartorius muscle and the anterior inferior iliac spine (AIIS) can be identified. After skin disinfection the needle is inserted placing the tip beneath the fascia iliaca at the lateral third of a line between the AIIS and pubic tubercle. Correct needle placement is confirmed by separation of the fascia iliaca from the iliopsoas muscle upon injection, with local anaesthetic spreading towards the FN medially and the iliac crest laterally.
  Interventions: Other: Infrainguinal Fascia Iliaca Block

INTERVENTIONS:
Other: Pericapsular nerve Group Block — Patients of study group will receive PENG block with 20 mL of 0,375% levobupivacaine with 4 mg of dexamethasone
  Arms: PENG block: Study group
Other: Infrainguinal Fascia Iliaca Block — Patients of control group will receive an infrainguinal fascia iliaca block with 30 mL of 0,25 % levobupivacaine with 4 mg of dexamethasone
  Arms: Infrainguinal fascia iliaca block: Control group

SUMMARY:
Pain management is a crucial aspect of the care of hip fracture patients. Patients with poorly controlled pain have an increased risk of delirium, long-term functional impairment, and remain hospitalized longer. Today, to relieve hip fracture pain, fascia iliaca block is routinely performed in the emergency department in addition to other pain medications administered by vein or by mouth. Several studies have questioned the analgesic efficacy of this block, suggesting the superiority of the newer PENG block. The purpose of this multicenter, randomized study is to compare the analgesic efficacy of PENG block versus fascia iliaca block, hypothesizing the superiority of the new approach over the gold standard. Participants will be blindly assigned in a 1:1 ratio to the study or control group, recruited from the Emergency Departments of IRCCS Policlinico San Matteo and Colchester Hospital (UK).

The main outcome is represented by the reduction of pain after the two blocks, measured as %SPID (percentage of "pain intensity difference"), a value derived from VAS scale measurements in the first hour post-procedure. Secondly, we will evaluate the proportion of patients with satisfactory pain control, the amount of opioids used and the safety profile of the two approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Capacity to understand the aim of the study, the potential benefits and side-effects of the procedures
* Capacity to provide consent
* Capacity to provide a self-assessment of pain using the written VAS Scale
* Confirmed radiological diagnosis of hip fractures (including subcapitate, transcervical, intertrochanteric and perthrocanteric fractures)
* Moderate or severe worst pain (visual analogue scale, VAS >40 mm) (at rest or dynamic)

Exclusion Criteria:

* Known hypersensitivity to local anaesthetics
* Confirmed radiological diagnosis of subtrochanteric or diaphyseal femur fractures
* Hemodynamic instability
* Known diagnosis of severe cognitive impairment
* Dementia and/or delirium (defined by a 4AT score ≥ 2)
* Lack of capacity to provide consent and to understand the aim of the study
* BMI>35
* Body weight < 40 Kg
* Prior hip surgery on the same fracture side
* Mild worst pain (visual analogue scale, VAS < 40 mm) (at rest or dynamic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Pain relief over the 60-minutes following either block measured as the percentage of summed pain-intensity difference (%SPID) | Outcome assessed within 60 minutes following the block (PENG or FIB)
  Pain relief over the 60-minutes following either block measured as the percentage of summed pain-intensity difference (%SPID) (derived from V AS measurement at T0-T1- T2-T3-T4 as described above)

SECONDARY OUTCOMES:
33% SPID 33% (33%SPID) | Outcome assessed within 60 minutes following the block (PENG or FIB)
  Number of patients who achieve a percentage of summed pain-intensity difference of 33% (33%SPID)
50%SPID | Outcome assessed within 60 minutes following the block (PENG or FIB)
  Number of patients who achieve a percentage of summed pain-intensity difference of 50% (50%SPID)
Quantity of opioids | Outcome assessed within 60 minutes following the block (PENG or FIB)
  Quantity of opioids (milligrams of morphine) administered in the first 60 minutes following either block
Adverse events | Outcome assessed within 60 minutes following the block (PENG or FIB)
  Occurrence of adverse events including nausea or vomiting, hypotension, respiratory depression (hypoxia or hypopnea), local anaesthetic toxicity syndrome (LAST syndrome) during ED stay (post-block). Adverse event will be described, and their incidence will be presented with 95% CI and compared with Fisher test.

CONTACTS AND LOCATIONS:
Overall Officials: Santi Di Pietro, MD, PhD, Principal Investigator — IRCCS San Matteo Foundation - University of Pavia
Locations (1):
- Emergency Department, IRCCS San Matteo University Hospital, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-05-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT05370586/Prot_001.pdf